CLINICAL TRIAL: NCT03206216
Title: Feasibility Study of New Method of Diagnostic and Prediction of Painful CIPN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Oliver Dorigo, Associate Professor of Obstetrics and Gynecology, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-40358; NCI-2017-01098 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GYN0006 (Other: OnCore)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Burning Pain; Impaired Balance; Malignant Ovarian Neoplasm; Numbness; Peripheral Neuropathy; Pain, Acute; Tingling
MeSH Terms: conditions — Pain; Ovarian Neoplasms; Hypesthesia; Peripheral Nervous System Diseases; Acute Pain; Paresthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A - Painful CIPN (Experimental): Participants with painful chemotherapy-induced peripheral neuropathy (CIPN) undergo Diode Laser fiber type Selective Stimulator (DLss) test over 30 minutes at 9 and 21 weeks after the first day of standard of care chemotherapy. A questionnaire is used to assess the level of pain after stimulation.
  Interventions: Diagnostic Test: Diode Laser fiber type Selective Stimulator (DLss)
- Group B - Painless CIPN (Active Comparator): Participants with painless chemotherapy-induced peripheral neuropathy (CIPN) undergo Diode Laser fiber type Selective Stimulator (DLss) test over 30 minutes at 9 and 21 weeks after the first day of standard of care chemotherapy. A questionnaire is used to assess the level of pain after stimulation.
  Interventions: Diagnostic Test: Diode Laser fiber type Selective Stimulator (DLss)

INTERVENTIONS:
Diagnostic Test: Diode Laser fiber type Selective Stimulator (DLss) — A laser device to assess pain sensitivity to stimulation
  Other Names: PNS

SUMMARY:
This clinical trial studies how well Diode laser fiber type Selective Stimulator (DLss) works in predicting pain development in patients with ovarian cancer who are receiving chemotherapy. Stimulating of the pain nerve fibers in the skin with laser light stimulation may help to predict whether a patient will develop painful peripheral neuropathy, correlate with the severity of neuropathy during and after chemotherapy treatment, and may help to explain the mechanisms of chemotherapy-induced neuropathic pain (CIPN).

DETAILED DESCRIPTION:
Laser stimulation, similar to what is being used in the DLss, has been used in pain clinics and research since 1975 as a diagnostic test for pain sensitivity. It is widely considered to be both useful and safe. Laser irradiation /stimulation simultaneously can activate either the heat-sensitive A-delta or C never fibers, with the difference in affected nerves being primarily on the basis of different pulse duration and different diameter of the simulation target. The laser for both type of simulation is set to 980 nanometers.

Laser irradiation intensity is measured as the milli-amperes (mA) required to generate that laser intensity. The pain sensitively of A-delta and C fibers are assessed by specific protocols (A-delta protocol: 60 millisecond duration, 980 nm stimuli, 1 mm diameter simulation target. C protocol: 2 second duration, 5 mm diameter simulation target).

Pain sensitivity is assessed as the ratio of painful laser intensity between the A-delta and C fibers (A-delta:C pain ratio).

Participants with ovarian cancer, with either painful (Group A) or painless (Group B) chemotherapy-induced peripheral neuropathy (CIPN), were to be assessed for pain sensitivity after 9 and 21 weeks of chemotherapy with Diode Laser fiber type Selective Stimulator (DLss). Both painful or painless CIPN are undesirable chemotherapy-induced side effects. The same testing protocol was used for these groups (ie, any difference between the groups would be attributed to differences in pain sensitivity between the groups). Patients would report the stimulation on a 0 to 100 scale, with 0 = no sensation; 10 = definite sensation; 0 to 40 = "painful"; and 100 = worst imaginable pain.

PRIMARY OBJECTIVES:

* Determine if there is a difference in the A-delta:C pain threshold ratio for patients with painful chemotherapy-induced peripheral neuropathy (CIPN) compared to patients with painless CIPN.
* Determine the A-delta:C ratio over time in patients with CIPN.

ELIGIBILITY:
INCLUSION CRITERIA

* Pathologically-proven ovarian cancer, or cancer of mullerian origin, that was or will be treated with a 1st-line taxane plus a platinum-based chemotherapy regimen.
* GROUP A (painful neuropathy group): Subjective symptoms of painful peripheral neuropathy (burning, stabbing, throbbing, painful tingling, aching in the fingers and/or toes) that is greater than or equal to 10 on a scale of 0 to 100 in the neuropathic pain questionnaire
* GROUP B (painless neuropathy group): Subjective symptoms of painless neuropathy (loss of sensation, worsening balance, strange sensation in fingers and/or toes) or no complaints related to neuropathy.
* Life expectancy of 6 months
* Ability to understand the study protocol, participate in testing, and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA

* Received prior chemotherapy for ovarian cancer or cancer of mullerian origin other than 1st-line treatment with a taxane + platinum based regimen.
* No concurrent investigational drugs.
* Received investigational drugs suspected to cause peripheral neuropathy.
* History of B12 deficiency
* History of neuropathy or numbness/tingling suspicious for neuropathy, prior to the first dose of chemotherapy for ovarian cancer
* Prior treatment for other cancers that included drugs known to cause neuropathy (including but are not limited to vinca-alkaloids, platinums, taxanes, bortizomib).
* Known peripheral vascular disease
* Chronic daily headache or headache for more than 14 days of the month
* Pain rated 50 or higher on a scale of 0 to 100, with 0 = no pain at all and 100 = worst pain imaginable.
* Pregnant or nursing
* HIV-positive
* Do not speak or read English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females equal to or greater than 18 years of age
Enrollment: 1 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Dorigo, MD, PhD, Study Chair — Stanford University; Seema Nagpal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A - Painful CIPN | Group B - Painless CIPN
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: No participants accrued to Group A Painful CIPN prior to study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Painful CIPN | Group B - Painless CIPN | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: A-delta:C Pain Threshold Ratio
Description: The "A-delta:C pain threshold ratio" is calculated based on the A-delta-fiber and C-fiber pain thresholds. The outcome was the difference in the A-delta:C pain ratio between the 9-week assessment and the 21-week assessment, to be reported as the mean with standard deviation for participant with painful CIPN (Group A) or painless CIPN (Group B).
Time Frame: Up to 24 weeks
Population: The only participant withdrew before the 21-week assessment. No outcome assessment is possible.
Arm/Group | Group A - Painful CIPN | Group B - Painless CIPN
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Correlation Between the "Adelta:C Pain Threshold Ratio" and Pain Development
Description: A Spearman correlation coefficient will be obtained for the A-delta:C pain threshold ratio as measured at 9 weeks (dependent variable) assessed against the presence or absence of pain (binary pain value) at 21 weeks (independent variable). The Spearman correlation coefficient will be obtained by logistic regression analysis.
Time Frame: Up to 24 weeks
Population: The only participant withdrew before the 21-week assessment. No outcome assessment is possible.
Arm/Group | Group A - Painful CIPN | Group B - Painless CIPN
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Description: No participants accrued to Group A Painful CIPN prior to study termination.
Arm/Group | Group A - Painful CIPN | Group B - Painless CIPN
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT03206216/Prot_SAP_000.pdf